CLINICAL TRIAL: NCT07059897
Title: Evaluatıon of the Effectiveness of the Video and Mobile Phone Application Prepared to Creat Awareness and Behavior ın Breast Cancer Screening
Brief Title: Effectiveness of a Video and Mobile App in Breast Cancer Screening Awareness
Acronym: Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Özlem BEKDEMİR AK (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Sponsor-Investigator, Özlem BEKDEMİR AK, Doctor-Midwife, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022/27; Project number: 36577 (Other Grant/Funding Number: İÜC-BAP)
Record Dates: First submitted 2025-06-12; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer Awareness
Keywords: animation video; MEKTUPmobilephone application; National Breast Cancer Screening Program in Turkey

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The study was conducted on 90 women aged 40-69 who had no symptoms of breast cancer. (Other): The research was done in 4 stages. The first phase (First encounter with cases/0th month); Informed Voluntary Consent Form (ANNEX-1), Individual Information Form (ANNEX-2), National Breast Cancer Screening Program Knowledge Test (Pre-test) (ANNEX-3) were applied. They were allowed to watch the animation video (ANNEX-4) via social media (Whatsapp).
  In the second phase (month 1); National Breast Cancer Screening Program Knowledge Test (Interim test) (ANNEX-3) was applied. They were asked to use the MEKTUP mobile phone application (ANNEX-5) by being trained.
  In the third stage (month 2); A reminder message was automatically sent to them to participate in breast cancer screenings with the MEKTUP mobile phone application (ANNEX-5)
  In the fourth stage (month 3); National Breast Cancer Screening Program Knowledge Test (Post-test) (ANNEX-3) and Research Evaluation Survey (ANNEX-6) were applied. A reminder message was sent with the MEKTUP mobile phone application (ANNEX-5).
  Interventions: Behavioral: Animation video and mobile phone application

INTERVENTIONS:
Behavioral: Animation video and mobile phone application — An animation video scenario and MEKTUP mobile phone application were prepared by the researchers in light of the literature, in line with the "National Breast Cancer Screening Program" and by taking expert opinions.

SUMMARY:
Introduction: Breast cancer is the most common type of cancer in women in the worldandinTurkey. It also ranks first in cancer-related deaths in women. Lack of awareness about thedisease, lack of information, late diagnosis and inadequate medical facilities cause anincreasein breast cancer incidence and mortality. Objective: To evaluate the effectiveness of a video and mobile phone application preparedtoraise awareness and turn breast cancerscreening into behavior in women aged 40-69 who do not have breast cancer symptoms.

Method: A quasi-experimental study based on design and comparison of pre test, midtest andpost test results of women in a single group. Data were collected via an online surveyandGoogle Play Store (to download the mobile phone application) between May 2023 andJanuary2024. The study was completed with 90 women. Data were collected using an individual information form, Breast Cancer Screening Program information test, animation video, Breast Cancer Screening Warning Program (MEKTUP) mobile phone application, and research evaluation survey.

DETAILED DESCRIPTION:
No study was found in Turkey on the combined use of animated videos and mobile phone applications to create awareness and behavioral changes for women to participate in breast cancer screening programs.

The research was conducted to evaluate the effectiveness of an animated video and mobile phone application prepared to raise awareness and turn it into behavior in asymptomatic women between the ages of 40-69 about performing BSE regularly every month, having BSE once a year, and having mammography once every two years.

Hypothesis₁: Watching an informative animated video about early screening program for breast cancer has a positive effect on the behaviors of women between the ages of 40-69 in terms of performing BSE, having CBE and having mammography.

Hypothesis₂: The reminder MEKTUP mobile phone application about early screening program for breast cancer has a positive effect on the behaviors of women between the ages of 40-69 in terms of performing BSE, having CBE and having mammography.

Hypothesis₃: Watching an animated video about early screening program for breast cancer and the reminder MEKTUP mobile phone application have a positive effect on the behaviors of women between the ages of 40-69 in terms of performing BSE, having CBE and having mammography.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 40-69
* The participant must live in Turkey
* Have internet access
* Being literate
* Having a smart phone and knowing how to use it
* Being a WhatsApp, Instagram or e-mail user
* No history of breast cancer
* No history of benign breast diseases such as cysts, fibroadenomas and hyperplasia in the breast
* No history of endometrial and/or ovarian cancer/cancer
* Not being visually or hearing impaired

Exclusion Criteria:

* Forms sent by the researcher not filled out or filled in incompletely
* Not watching the video
* Not using the mobile phone application regularly
* Women who regularly participate in breast cancer screening programs

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Woman
Enrollment: 90 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
National Breast Cancer Screening Program Knowledge Test (At the first stage (first encounter with cases/month 0)) | first encounter with cases/month 0
  After the informed written consent was received from the women who agreed to participate in the research, the Descriptive Information Form prepared by the researchers and the National Breast Cancer Screening Program Knowledge Test were applied as the "Pre-Test" via e-mail or social media.
  The Descriptive Information Form contains 17 questions about age, marital status, education level, employment, income status, last menstrual period, smoking, a family history of breast cancer, and breast cancer early screening program.
  National Breast Cancer Screening Program Knowledge Test: This test was prepared using the literature and the National Breast Cancer Screening Program .The test includes a total of 20 questions, with 10 correct and 10 incorrect answers. If an individual answers all questions correctly, they score 20 points.
National Breast Cancer Screening Program Knowledge Test (At the second stage (month 1)) | month 1
  The National Breast Cancer Screening Program Knowledge Test was applied to the women who watched the animated video a second time, one month later, as the "Interim Test" via. Immediately after the interim test, the participants were interviewed and asked to download the MEKTUP mobile phone application from the Google Play Store and register. The mentioned video was sent to the participants via WhatsApp.
  Animated Video: An animated video scenario was prepared by reviewing the literature and based on the "National Breast Cancer Screening Program". Written expert opinions were received on both the video design and information content. Three characters (a mother, a daughter, and a doctor) were included in the animation design. In the scenario, the doctor provided information on how, when, and where to perform BSE, undergo CBE, and have mammography, and breast cancer symptoms. (Animated video)
National Breast Cancer Screening Program Knowledge Test (At the second stage (month 1)) | month 1
  The National Breast Cancer Screening Program Knowledge Test was applied to the women who watched the animated videoa second time, one month later, as the "Interim Test" via. Immediately after the interim test, the participants were interviewed and asked to download the MEKTUP mobile phone application from the Google Play Store and register. The mentioned video was sent to the participants via WhatsApp.
  The Breast Cancer Screening Warning Program (MEKTUP) mobile phone application, designed by the researchers in line with the "National Breast Cancer Screening Program" and having a reminder feature, was employed as a data collection tool. The mobile phone application automatically sent reminder messages in the "Reminder" section to menstruating women, according to the date of their last menstruation, and to non-menstruating women, according to a date they determined, to perform BSE once a month, to undergo CBE once a year, and to have mammography once every two years.
the MEKTUP mobile phone application (At the third stage) | month 2
  Reminder messages were automatically sent to women concerning breast cancer screening follow-ups via the MEKTUP mobile phone application according to their last menstrual date or the dates they provided.
the Research Evaluation Survey (At the fourth stage) | month 3
  The National Breast Cancer Screening Program Knowledge Test applied to women at the first meeting was filled out for the third time as the "Post-Test." Furthermore, the effects of the animated video and the MEKTUP mobile phone application on women's knowledge about the breast cancer screening program and their behaviors were evaluated using the Research Evaluation Survey.
  Research Evaluation Survey:The said survey comprises six questions about women's status of participating in breast cancer screenings and the effects of the animated video and the MEKTUP (LETTER) mobile phone application on their participation in breast cancer screenings at the fourth research stage.

CONTACTS AND LOCATIONS:
Overall Officials: Nuran GENÇTÜRK Associate Professor, Study Director — İstanbul University-Cerrahpasa
Locations (1):
- İstanbul Üniversitesi-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No